CLINICAL TRIAL: NCT05567874
Title: Proportion of Nosocomial COVID-19 Infections in Patients Hospitalized at the Metz-Thionville Regional Hospital in 2021
Brief Title: Nosocomial COVID-19 Infections in Patients Hospitalized at the Metz-Thionville Regional Hospital in 2021
Acronym: COVIDIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-09Obs-CHRMT
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-10

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV 2 infected patients hospitalized at CHR Metz-Thionville in 2021 during the first period: SARS-CoV 2 infected patients hospitalized at CHR Metz-Thionville in April 2021
  Interventions: Other: Nosocomial SARS-COV 2 Infection proportion
- SARS-CoV 2 infected patients hospitalized at CHR Metz-Thionville in 2021 during the second period: SARS-CoV 2 infected patients hospitalized at CHR Metz-Thionville from June to September 2021
  Interventions: Other: Nosocomial SARS-COV 2 Infection proportion
- SARS-CoV 2 infected patients hospitalized at CHR Metz-Thionville in 2021 during the third period: SARS-CoV 2 infected patients hospitalized at CHR Metz-Thionville in December 2021
  Interventions: Other: Nosocomial SARS-COV 2 Infection proportion

INTERVENTIONS:
Other: Nosocomial SARS-COV 2 Infection proportion — Proportion of Nosocomial SARS-COV 2 Infections in Patients Hospitalized at the Metz-Thionville Regional Hospital in 2021

SUMMARY:
The rate of nosocomial SARS-CoV2 infections found in the different studies since the beginning of the pandemic is very variable (<1% in hospitals in the USA to about 20% in a British hospital). Mortality related to these nosocomial SARS-CoV2 infections is higher than in the general population. The risk factors identified for this nosocomial acquisition are multiple. We were confronted with nosocomial acquisitions and cluster situations in the services, without exhaustive data to measure these phenomena, and we lacked data to consider areas for improvement.

The objectives of this study are to determine the proportion of nosocomial SARS COV 2 infections in the total number of patients hospitalized with a Covid-19 infection at the CHR Metz-Thionville in 2021, and to describe the characteristics of this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised at the CHR Metz-Thionville in medicine, surgery and obstetrics (MCO) or geriatric follow-up and rehabilitation care (SSR) units, in 2021 for a Covid-19 infection defined by the existence of a positive PCR result for SARS-CoV2 during the stay, or by the existence of an ICD10 code for COVID in the PMSI data of the health care establishment

Exclusion Criteria:

* Opposition to participate in the study after reading the patient information note.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with Covid-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of hospital-acquired infections in patients hospitalised with a covid-19 infection | up to 8 months after the third COVID-19 wave
  Several elements are taken into account: a) the time between entry into the establishment and the first positive SARS COV 2 PCR, b) the time between entry into the establishment and the appearance of the most frequent symptoms (fever, cough), if present in the patient, in the seven days preceding the first positive SARS COV 2 PCR, c) the existence of an epidemiological link with other infected patients, via contact in a double room with another case, and/or via hospitalisation in a department concerned by a cluster situation according to the Santé Publique France definition of May 2020 (identified on the basis of monitoring and surveillance data from the hygiene department).

SECONDARY OUTCOMES:
Description of the nosocomial infected population | up to 8 months after the third COVID-19 wave
  age, sex, hospital unit care, outcomes of stay, vaccination status, associated conditions (comorbidities according to Charlson score, obesity, pregnancy), existence of screening on admission, time to acquisition of nosocomial infection, number of negative SARS-COV 2 PCRs in the institution before the first positive PCR, type of variant, presence of symptoms (cough, fever), stay in a double room in the 14 days prior to infection, cluster status in the ward, length of stay after infection.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu LLORENS, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France